CLINICAL TRIAL: NCT01782547
Title: Telehealth Intervention for Youth With Type 1 Diabetes
Brief Title: Telehealth Intervention for Youth With T1DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Erinn T. Rhodes, Director of Endocrinology Healthcare Research and Quality, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00006175
Record Dates: First submitted 2013-01-28; First posted 2013-02-04 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes mellitus; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telehealth Intervention (Experimental): Telehealth intervention - 6 months
  Interventions: Behavioral: Telehealth Intervention
- Usual care (Active Comparator): Usual care control with comparable frequency of contact
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Telehealth Intervention — Monthly videoconference with diabetes nurse educator; Monthly videoconference with social worker; Diabetes action plan;
  Arms: Telehealth Intervention
Other: Usual Care — Standard diabetes care- typically a visit with a diabetes health care provider every 3 months and referrals to a dietitian or mental health specialist as deemed appropriate; Study participation reminder cards twice per month
  Arms: Usual care

SUMMARY:
Hospitalization of youth with established diabetes is both costly and frequently preventable. Poor glycemic control is a risk factor for hospitalization and is also associated with adolescent age and lower socioeconomic status. This is a randomized, controlled trial for high-risk adolescent youth with T1DM and suboptimal glycemic control with an intervention arm and usual care control arm matched for frequency of contacts. There will be 110 subjects with T1DM and HbA1c>8%, aged 13 to 17 years, recruited from the Diabetes Program at Boston Children's Hospital and followed for 6 months. The intervention will be implemented by a diabetes nurse educator and social worker, who will each have monthly contact with the adolescent and a parent/guardian through a telehealth (videoconference) visit. Care will be guided by a diabetes action plan. Telehealth interventions have been utilized successfully in both adults and youth with diabetes. They facilitate frequent contact with the care team allowing barriers to adherence to be addressed, education to be reinforced, care plans to be updated, and diabetes-specific family support to be provided.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 to 17 years
* Type 1 diabetes for ≥1 year
* HbA1c>8%
* Able to speak and read English (Child)
* Able to speak and read English (Parent)
* Parent agrees to participate
* Parent and child each have email addresses

Exclusion Criteria:

* Plan to transition diabetes care to a center other than Boston Children's Hospital
* No visit to Boston Children's Hospital Diabetes Program in year prior to recruitment
* Current participation in another diabetes-related study with an intervention
* Living with or related to another study participant
* Significant psychopathology or medical illness that would limit the subject's ability to provide assent and/or participate in the study procedures as determined by the PI.
* No internet access

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | baseline and 6 months
  Change in hemoglobin A1c over 6 months

SECONDARY OUTCOMES:
% patients meeting ADA HbA1c target | At 6 months
  proportion of patients meeting the American Diabetes Association target for optimal glycemic control in this age group, which is <7.5%
Diabetes-related adverse events | Up to 6 months
  number of diabetes-related hospitalizations, ED visits, and episodes of severe hypoglycemia
Change in Diabetes self-efficacy | Baseline and 6 months
  change over 6 months assessed by questionnaire
Change in Adherence to diabetes self-management | Baseline and 6 months
  change over 6 months assessed by questionnaire
Change in competence with diabetes skills | Baseline and 6 months
  change over 6 months assessed by questionnaire
Change in Health related quality of life | Baseline and 6 months
  change over 6 months assessed by questionnaire
Change in Diabetes Knowledge | Baseline and 6 months
  Change over 6 months assessed by questionnaire

OTHER OUTCOMES:
Direct medical costs | Up to 6 months
  Direct medical costs include planned intervention costs and medical costs that are expected to change as a result of the intervention.
Change in diabetes-related family conflict | Baseline and 6 months
  assessed by questionnaire
Change in family responsibility for diabetes tasks | Baseline and 6 months
  assessed by questionnaire
Telehealth intervention satisfaction | At 6 months
  satisfaction, engagement, visit characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Erinn T Rhodes, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States